CLINICAL TRIAL: NCT06333340
Title: Comparative Efficacy of Carbetocin and Oxytocin in Parturients at Risk of Atonic Postpartum Hemorrhage Undergoing Elective Cesarean Delivery: a Randomized Controlled Trial
Brief Title: Comparative Efficacy of Carbetocin and Oxytocin in Parturients at Risk of Atonic Postpartum Hemorrhage Undergoing Elective Cesarean Delivery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24-03
Record Dates: First submitted 2024-03-15; First posted 2024-03-27 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Post Partum Hemorrhage
Keywords: oxytocin; carbetocin; cesarean delivery; pregnancy
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin; carbetocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin 5IU (Active Comparator): IV oxytocin 5 IU diluted in 10 mL normal saline over 1 min followed by continuous infusion of 250 mIU/min over 4 hours.
  Interventions: Drug: Oxytocin
- Carbetocin 100mcg (Active Comparator): IV carbetocin 100 mcg diluted in 10 mL normal saline over 1 min followed by placebo infusion for 4 hours after the delivery of the fetus.
  Interventions: Drug: Carbetocin

INTERVENTIONS:
Drug: Oxytocin — Patient is given oxytocin 5 IU diluted in 10 mL normal saline, administered intravenously over 1 min, followed by continuous infusion of 250 mIU/min over 4 hours.
  Other Names: Pitocin
  Arms: Oxytocin 5IU
Drug: Carbetocin — Patient is given carbetocin 100 mcg diluted in 10 mL normal saline, administered intravenously over 1 min, followed by placebo infusion for 4 hours.
  Other Names: Duratocin
  Arms: Carbetocin 100mcg

SUMMARY:
The goal of this study is to compare 2 medications that are commonly used to prevent excess uterine bleeding (postpartum hemorrhage, or PPH) following cesarean delivery (CD), oxytocin and carbetocin. Most of the trials evaluating the preventative role of oxytocin and carbetocin after CD have focused on patient with low-risk of PPH.

This trial will focus on patients that are at increased risk of PPH, with risk factors such as: multiple gestation (twins, or more multiples), large baby, polyhydramnios (excess amniotic fluid), history of PPH, body mass index greater than 40, diabetes mellitus, hypertension, and placenta previa.

The investigators hypothesize that carbetocin would be more effective than an oxytocin regimen in reducing the risk of PPH in patients undergoing CD with any of the biological high-risk factors.

DETAILED DESCRIPTION:
Postpartum hemorrhage (PPH) is a potentially life-threatening complication and one of the leading causes of maternal mortality. It has been estimated that one in every five maternal deaths occurs due to PPH globally. Primary PPH is predominantly caused by uterine atony or inadequate contraction of the uterus after childbirth. Active management of the third stage of labor involves prophylactic administration of a uterotonic agent before delivery of the placenta, as well as delayed cord clamping and controlled traction of the umbilical cord. The uterotonic administration remains the most essential component in terms of preventing PPH.

Oxytocin, a synthetic pituitary hormone, is the most commonly used first-line uterotonic drug. However, because of the short half-life (3-17 min), a continuous intravenous infusion is necessary to maintain uterotonic activity. Carbetocin is a synthetic oxytocin analog that binds with a similar affinity to the oxytocin receptors in the myometrium. Carbetocin produces stronger and more sustained action compared to oxytocin and has a longer half-life than oxytocin, thus reducing the requirement for an infusion after the initial dose. Recently published guidelines from the Society of Obstetrics and Gynecology (SOGC) have stated that Carbetocin should be considered as a first-line agent for the prevention of PPH after cesarean delivery (CD). The international consensus statement on the use of uterotonic agents has also recommended carbetocin as an alternative to oxytocin infusion during CD due to its longer duration of action.

Trials comparing carbetocin with oxytocin in CD have shown mixed results on superiority of carbetocin over oxytocin for the need for additional uterotonics and amount of blood loss, however, no significant effect on blood loss >1000 ml could be found. Most of the trials evaluating the prophylactic role of oxytocin and carbetocin after CD have focused on the low-risk PPH population. The incidence of biological risk factors for uterine atony such as multiple gestation (due to assisted reproductive techniques), and obesity has progressively increased in developed countries. There is still a lack of high-quality trials on the efficacy of carbetocin in high-risk parturients undergoing CD.

In this study, the investigators aim to compare the efficacy of carbetocin 100 mcg with oxytocin 5 IU bolus followed by continuous infusion of 250 mIU/min over 4 hours at elective CD in parturients with risk factors for uterine atony.

The comparative data is still lacking for both the agents as first-line uterotonics for patients having a high risk for uterine atony undergoing cesarean delivery. The result of this trial regarding the relative uterotonic efficacy and safety of the standardized prophylactic doses of both agents (carbetocin and oxytocin) will form the evidence base for future guidelines in high-risk parturients.

ELIGIBILITY:
Inclusion criteria - Any one or more of the risk factors for uterine atony:

* Overdistended uterus due to:

  * Polyhydramnios (amniotic fluid index >24 cm)
  * Fetal macrosomia reported on prenatal ultrasound >90th centile or > 4000 gm
  * Multiple gestation
* History of uterine atony/PPH (documented with blood loss of >1000 ml, blood transfusion, use surgical methods such as Bakri balloon, B-Lynch sutures, uterine artery ligation or embolization)
* Obesity with body mass index (BMI) >40 kg/m2
* Diabetes mellitus on treatment
* Preeclampsia on treatment
* Placenta previa

Exclusion criteria:

* Valvular heart disease, arrhythmias, or heart failure
* Placenta accreta spectrum
* Bleeding disorder
* Anemia (<100 g/dl)
* Allergy or sensitivity to oxytocin or carbetocin

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of parturients requiring additional uterotonic agents intraoperatively | 90 minutes
  The proportion of patients who are administered additional uterotonic agents intraoperatively will be divided by the total number of patients assigned to the same treatment arm, for each of the 2 groups: oxytocin and carbetocin.

SECONDARY OUTCOMES:
Uterine Tone 3 minutes | 3 minutes
  The intensity of uterine tone as evaluated by palpation of the uterus by the obstetrician at 3 minutes, from the completion of delivery of the drug, utilizing a verbal numeric rating scale of 0-10.
Uterine Tone 5 minutes | 5 minutes
  The intensity of uterine tone as evaluated by palpation of the uterus by the obstetrician at 5 minutes, from the completion of delivery of the drug, utilizing a verbal numeric rating scale of 0-10.
Uterine Tone 10 minutes | 10 minutes
  The intensity of uterine tone as evaluated by palpation of the uterus by the obstetrician at 10 minutes, from the completion of delivery of the drug, utilizing a verbal numeric rating scale of 0-10.
Calculated blood loss (CBL) | 24 hours
  Blood loss will be calculated through the difference in hematocrit values assessed prior to and at the end of 24 hours after the cesarean section.
Semi-quantitative blood loss (SQBL) | 2 hours
  Blood loss measured in the operating room by volume (ml)
Presence of blood transfusion | 24 hours
  Number of units of blood product administered post-delivery
Number of patients with ICU admission | 24 hours
  Admission to the intensive care unit for bleeding post partum
Number of patients with conservative surgical methods to manage post partum hemorrhage | 2 hours
  Bakri balloon/B-Lynch sutures used intraoperatively
Number of patients with radiological methods used to manage post partum hemorrhage | 2 hours
  Uterine artery embolization used intraoperatively.
Number of patients with surgical post partum hemorrhage management measures | 2 hours
  Re-exploration for bleeding/uterine artery ligation/hysterectomy
Number of patients with hypotension defined as systolic blood pressure less than 80% of baseline | 2 hours
  Systolic blood pressure < 80% of baseline, at any time during surgery
Number of patients with hypertension defined as systolic blood pressure greater than 120% of baseline | 2 hours
  Systolic blood pressure > 120% of baseline, at any time during surgery
Number of patients with tachycardia defined as heart rate greater than 130% of baseline | 2 hours
  Heart rate > 130% of baseline, at any time during surgery
Number of patients with bradycardia defined as heart rate less than 70% of baseline | 2 hours
  Heart rate < 70% of baseline, at any time during surgery
Presence of ventricular tachycardia: ECG | 2 hours
  Presence of ventricular tachycardia as recorded by ECG, at any time during surgery
Presence of atrial fibrillation: ECG | 2 hours
  Presence of atrial fibrillation as recorded by ECG, at any time during surgery
Presence of atrial flutter: ECG | 2 hours
  Presence of atrial flutter as recorded by ECG, at any time during surgery
Presence of nausea: questionnaire | 2 hours
  The presence of nausea at any time during surgery, as reported by the patient
Presence of vomiting: questionnaire | 2 hours
  The presence of vomiting at any time during surgery, as reported by the patient
Number of patients with chest pain: questionnaire | 2 hours
  Any presence of chest pain, at any time during surgery, as reported by the patient
Number of patients with shortness of breath: questionnaire | 2 hours
  Any presence of shortness of breath, at any time during surgery, as reported by the patient.
Number of patients with headache: questionnaire | 2 hours
  Any presence of headache, at any time during surgery, as reported by the patient.
Number of patients with flushing: questionnaire | 2 hours
  Any presence of flushing, at any time during surgery.
Additional uterotonics administered up to 24 hours post delivery: questionnaire | 24 hours
  Were any additional uterotonics administered up to 24 hours post delivery: yes or no Detailed description of any medication and dosage recorded.
Obstetric Quality of Recovery-10 (ObsQoR-10) score 24 hours | 24 hours
  ObsQoR-10 score at 24 hours. There are 10 questions, and the results are tabulated out of 100. The higher the overall score out of 100, the better quality of recovery a patient is experiencing.

CONTACTS AND LOCATIONS:
Overall Officials: Mrinalini Balki, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No